CLINICAL TRIAL: NCT01172730
Title: Use of Ultrasound to Measure Depth of Thoracic Epidural Space Compared With Blind Technique
Brief Title: The Use of Ultrasound to Measure Depth of Thoracic Epidural Space
Status: Completed | Type: Observational
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Issam Khayata, Study Principle Investigator, University of Massachusetts, Worcester
Other Study IDs: 13495
Record Dates: First submitted 2010-05-24; First posted 2010-07-30 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Post Operative Trauma; Acute Pain
Keywords: Post operative pain; thoracic epidural; acute pain; Ultrasound scanning of the thoracic spine
MeSH Terms: conditions — Acute Pain; Pain, Postoperative | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ultrasound scanning
  Interventions: Device: Ultrasound scanning

INTERVENTIONS:
Device: Ultrasound scanning — Ultrasound scanning is used to define needle insertion point and depth of epidural space.
  Other Names: LogicE GE portable ultrasound machine

SUMMARY:
The purpose of the study is to evaluate the use of ultrasound scanning of the thoracic spine to define the point of insertion and the depth of the epidural space compared to the blind technique.

The study hypothesis is the use of Ultrasound will improve the success rate of epidural placement and may also decrease the rate of complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years and older having a thoracic epidural catheter
* Both male and female patients.

Exclusion Criteria:

* Pediatric population < 18 years of age
* Pregnancy
* Prisoners
* Absolute Contraindication to thoracic epidural placement severe scoliosis or deformity,
* Patients with previous spine surgery or hardware implanted at level of epidural placement,
* Anticipated ventilation postoperatively for a period more that 24 hrs
* Lack of patient consent to enroll in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having a thoracic epidural catheter for post operative pain
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2010-05; Primary Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
The success rate of epidural catheter to control pain | post operative day # 1

SECONDARY OUTCOMES:
The complication rate from epidural catheter placement. | Immediate complications 24 hrs after

CONTACTS AND LOCATIONS:
Overall Officials: Issam Khayata, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- UMass Memorial Medical Center, Worcester, Massachusetts, United States